CLINICAL TRIAL: NCT01089712
Title: Management Practices and the Risk of Infection Following Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: GCO 08-1078-00005; 5U01HL088942 (NIH); 5U1HL088942-02; 694 (Other: Ct Surgery Network Research Group)
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Cardiac Surgery; Infection, Postoperative Wound; Postoperative Wound Infection; Infections, Nosocomial; Management Practices
Keywords: Infection; Cardiac Surgery; Post Operative Cardiac Surgery Infection; Management Practices
MeSH Terms: conditions — Surgical Wound Infection; Cross Infection; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients undergoing cardiac surgery: The patient population for this study consists of all patients undergoing cardiac surgical interventions. All patients who meet the eligibility criteria may be included in the study regardless of gender, race or ethnicity.

SUMMARY:
The purpose of the study is to determine the best ways to prevent infections after heart surgery. Participation in the study will last at most 3 months after heart surgery. The study will only collect information about the care patients receive during the planned surgery. No new testing or procedures will be done. Patients will receive only the tests or procedures the doctor already has planned. This kind of study is an observational study, because all that is planned to do is observe the care patients receive and how well they do during treatment. The information collected should help to improve the quality of surgical care in the future.

DETAILED DESCRIPTION:
Hospital-acquired infections represent the main non-cardiac complication after heart surgery. They are associated with substantial morbidity and higher mortality, as they often require prolonged hospitalization and additional surgery. The proportion of cardiac surgery patients at high-risk for infection is increasing because of the increased prevalence of co-morbid conditions such as obesity and diabetes mellitus in the general (and especially the elderly) population.

In addition to increased morbidity and mortality, infectious complications also result in greater economic burden. A past study estimated that the incremental cost of treating Medicare beneficiaries who suffered from septicemia after coronary artery bypass grafting (CABG) to be $59,204. These patients stayed in the hospital 21.3 days longer than those who did not experience any serious adverse events. Of great relevance to treating hospitals, the Centers for Medicare and Medicaid Services (CMS) announced in the fall of 2007 that they would no longer pay for care related to preventable complications. CMS specifically mentioned excluding reimbursements for mediastinitis after CABG, and catheter associated infections. Thus, there is a crucial need to identify variables that mitigate infections post cardiac surgery and to develop effective preventative treatment strategies.

Prior studies have examined the relationship between patient baseline (preoperative) characteristics (e.g., co-morbid conditions) and hospital-acquired infections post cardiac surgery. The STS database, for example, has led to the identification of predictive factors of post-operative CABG infections. Much of the variations in outcomes seen at different institutions, however, cannot be explained by differences in preoperative patient characteristics alone. How care is delivered also plays an essential role in determining infection rates and is therefore likely to explain some of the differences in these rates observed at different institutions. The literature has not sufficiently examined the relationship between treatment/management practices (e.g., line management, ventilator management, etc) and postoperative infection risk. In this study we seek to better understand management practices that put patients at high risk for infections post-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for cardiac surgical interventions
* Age ≥ 18 years

Exclusion Criteria:

* Active systemic infection at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing cardiac surgical interventions at the 10 CT Surgery Network institutions
Sampling Method: Non-Probability Sample
Enrollment: 5158 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be major infection within 60 days of index cardiac surgical intervention. | 60 Days

SECONDARY OUTCOMES:
Major infection after surgery during the operative admission or within 30 days after discharge when associated with readmission. | 30 Days
Other infections within 60 days of index cardiac surgical intervention; Superficial incisional surgical site infection (primary/secondary); Symptomatic urinary tract infection; Asymptomatic bacteriuria | 60 Days
Non-infection adverse events within 60 days of index cardiac surgical intervention; Neurologic Dysfunction; Transient ischemic attack; cerebrovascular accident (ischemic or hemorrhagic stroke); Myocardial infarction | 60 Days
Re-operation within 60 days of index cardiac surgical intervention | 60 Days
Survival, All-cause mortality, Hospitalizations, Economic Measures | 60 Days

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Gardner, MD, Study Chair — Christiana Care Health Services; Patrick O'Gara, MD, Study Chair — Brigham and Women's Hospital; Annetine Gelijns, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (10):
- United States (9):
  - Emory University, Atlanta, Georgia
  - NIH Heart Center at Suburban Hospital, Bethesda, Maryland
  - Columbia University Medical Center, New York, New York
  - Montefiore Einstein Heart Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - East Carolina Heart Institute, Greenville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Greco G, Shi W, Michler RE, Meltzer DO, Ailawadi G, Hohmann SF, Thourani VH, Argenziano M, Alexander JH, Sankovic K, Gupta L, Blackstone EH, Acker MA, Russo MJ, Lee A, Burks SG, Gelijns AC, Bagiella E, Moskowitz AJ, Gardner TJ. Costs associated with health care-associated infections in cardiac surgery. J Am Coll Cardiol. 2015 Jan 6;65(1):15-23. doi: 10.1016/j.jacc.2014.09.079. PMID 25572505
- [Derived] Gelijns AC, Moskowitz AJ, Acker MA, Argenziano M, Geller NL, Puskas JD, Perrault LP, Smith PK, Kron IL, Michler RE, Miller MA, Gardner TJ, Ascheim DD, Ailawadi G, Lackner P, Goldsmith LA, Robichaud S, Miller RA, Rose EA, Ferguson TB Jr, Horvath KA, Moquete EG, Parides MK, Bagiella E, O'Gara PT, Blackstone EH; Cardiothoracic Surgical Trials Network (CTSN). Management practices and major infections after cardiac surgery. J Am Coll Cardiol. 2014 Jul 29;64(4):372-81. doi: 10.1016/j.jacc.2014.04.052. PMID 25060372
- See also: Cardiothoracic Surgical Trials Network — http://www.ctsurgerynet.org